CLINICAL TRIAL: NCT04948203
Title: SECOVID: A Multi-center, Randomized, Dose-ranging Parallel-group Trial Assessing the Efficacy of Sirolimus in Hospitalized Patients With COVID-19 Pneumonia for the Prevention of Post-COVID Fibrosis
Brief Title: Assessing the Efficacy of Sirolimus in Patients With COVID-19 Pneumonia for Prevention of Post-COVID Fibrosis
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB21-0400
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Fibrosis; COVID-19 Pneumonia; Long COVID
Keywords: SECOVID; Sirolimus; Rapamune; Post-COVID Fibrosis; PASC
MeSH Terms: conditions — Pulmonary Fibrosis; Post-Acute COVID-19 Syndrome | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sirolimus 0.5mg (Active Comparator): Subject will take Sirolimus 0.5mg orally daily for 14 days.
  Interventions: Drug: Sirolimus
- Sirolimus 1mg (Active Comparator): Subject will take Sirolimus 1mg orally daily for 14 days.
  Interventions: Drug: Sirolimus
- Sirolimus 2mg (Active Comparator): Subject will take Sirolimus 2mg orally daily for 14 days.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Triangular-shaped tablet
  Other Names: RAPAMUNE

SUMMARY:
The primary purpose of this study is to determine whether the drug sirolimus reduces the likelihood of developing of pulmonary fibrosis in patients who are hospitalized with COVID-19 pneumonia.

DETAILED DESCRIPTION:
Hospitalized patients with a diagnosis of COVID-19 pneumonia will be referred to the study team for potential recruitment. Initial screening will take place using the existing medical record and in collaboration with the treating team. The study consists of 3 randomly assigned arms of varying dosages of the study drug

All procedures, with the exception of drug dosing and option sample analysis, align with the subject's standard of care. Prior to initiating study drug, the subject's standard of care labs, imaging and oxygen requirements will be reviewed.

Sirolimus will be administered as an oral medication. Subjects who are discharged prior to receiving 14 days of study drug will be provided with enough study drug to finish at home.

On-study evaluation includes measurement of vital signs and laboratory studies before and after a patient has received sirolimus while inpatient. As part of routine care, subjects will be seen daily while in the hospital and will be monitored through blood tests for general health as well as renal function. Vital signs will be monitored daily while in the hospital, physical exams, assessment of COVID-19, and CT scans or chest x-rays as necessary for routine care.

Subjects will return to clinic at 12 weeks for routine lab work and imaging as a part of study follow-up and will be assessed for pulmonary fibrosis at this time.

Additionally, University of Chicago Medicine patients will have the option to allow investigators to use leftovers from tubes of blood drawn for clinical tests that would otherwise be discarded. This will apply to any blood collected during that respective hospital stay as well as up to 1 year after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Approval from the patient's primary inpatient service
* Hospitalized
* Diagnosed with COVID-19 pneumonia
* Positive test for active SARS-CoV-2 infection
* Requiring supplemental oxygen ≥ 5LNC or ≥ 40% FiO2.
* Chest computed tomography (CT) at admission with < 10% pulmonary fibrosis
* Ability to provide written informed consent on the part of the subject or, in the absence of decisional capacity of the subject, an appropriate surrogate (e.g. a legally authorized representative).

Exclusion Criteria:

* Known diagnosis of previous pulmonary fibrosis or an interstitial lung disease.
* Clinical features or known diagnosis of malignancy or active non-COVID-19 infection, including untreated latent tuberculosis.
* History of unstable or deteriorating cardiac disease (including myocardial infarction, coronary artery bypass surgery or angioplasty within the past 6 months, congestive heart failure requiring hospitalization within the past 6 months, or uncontrolled arrhythmia.
* Known history of hypersensitivity to sirolimus.
* History of unstable or deteriorating neurologic disease (including TIAs or stroke).
* Pregnant or lactating females. Females of child bearing potential are required to have a negative pregnancy test prior to treatment and practice abstinence or prevent pregnancy by at least a barrier method of birth control.
* Investigational therapy for any indication within 28 days prior to treatment.
* Current treatment with any drugs that are strong inhibitors of CYP3A4.
* Tofacitinib
* Clarithromycin
* Telithromycin
* Nefazodone
* Itraconazole
* Ketoconazole
* Atazanavir
* Darunavir
* Indinavir
* Lopinavir
* Nelfinavir
* Ritonavir
* Saquinavir
* Tipranavir.
* Inability or unwillingness to comply with the requirements for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Pulmonary Fibrosis as evidenced by CT scan | 12 Weeks
  Number of patients with >10% pulmonary fibrosis on chest CT

SECONDARY OUTCOMES:
10% Threshold for Pulmonary Fibrosis evidenced by CT scan | 12 Weeks
  Number of patients with >10% pulmonary fibrosis on chest CT
Qualitative Fibrotic markers on chest CT | 12 Weeks
  Number of patients with the presence or absence of chest CT imaging markers of fibrosis
Quantitative Fibrosis Score on chest CT | 12 Weeks
  Quantitative Fibrosis Score on chest CT
Duration of Increased Supplemental Oxygen from Baseline | 84 Days
  Number of days over which the participant requires supplemental oxygen in excess over baseline supplemental oxygen requirement.
Pulmonary Function Test impairment | 12 Weeks
  Number of subjects with the presence of abnormal indices of lung function tests

OTHER OUTCOMES:
Safety - Rate of Liver Function Test abnormalities | 12 Weeks
  Number of patients in a study arm who develop severe impairment of liver function tests exceeding three times the upper limit of normal

CONTACTS AND LOCATIONS:
Overall Officials: Ayodeji Adegunsoye, MD, MS, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No